CLINICAL TRIAL: NCT06308991
Title: The Effect of Yakson and Gentle Touch Method on Pain, Comfort and Physiological Parameters in Preterm Infants During Endotracheal Aspiration
Brief Title: Effect of Touch Methods in Preterm Infants During Endotracheal Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Sadiye Dur, Assistant Professor, Izmir Democracy University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IDU-SBF-SD-01
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Endotracheal Aspiration
Keywords: Therapeutic Touch; Pain; Preterm Infant
MeSH Terms: conditions — Pain; Premature Birth

STUDY DESIGN:
Intervention Model Description: The order of the 2 different touching methods and routine care practices to be applied to the infants in the research group was determined by randomized method and 3 groups were created. Considering the order of application in each group, it was decided which touch method and routine care would be applied to the infants. Both touch techniques and routine care practices were applied once to each infant.
  Group 1: Yakson touch, Routine care, Gentle HumanTouch Group 2: Routine care, Gentle HumanTouch, Yakson touch Group 3: Gentle HumanTouch, Yakson touch, Routine care
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yakson touch (Experimental): The Yakson method continued for 15 minutes with steady touch (5 minutes), compassionate caressing (5 minutes), and repetition of steady touch (5 minutes). In the Yakson touch method, the palms of the practitioner and all fingers were kept in close contact so that the infants did not feel pressure.
  1. Steady touch (5 minutes): One hand rested on the chest and abdomen of the preterm infant, while the other hand supported the back and hip of the preterm infant.
  2. Compassionate Caress (5 minutes): In the same hand position, the practitioner repeated caressing and resting for 5 minutes: Caress (1 minute), rest (30 seconds), caress (1 minute), rest (30 seconds), and caress (2 minutes). The practitioner caressed the infants' chest and belly with a 1 cm diameter clockwise circular movement every 10 seconds.
  3. Steady touch (5 minutes): The practitioner followed the steady touch procedure as previously described.
  Interventions: Other: Yakson touch
- Gentle Human Touch (Experimental): While the practitioner placed one hand on the crown of the preterm infant on the eyebrow line with the fingertip touch for 15 minutes, the other hand was placed on the lower abdomen covering the waist and hip of the infant.
  Interventions: Other: Gentle Human Touch
- Routine Care (Other): All infants in the control, Yakson, and GHT groups were applied swaddling as the routine practice of the clinic before and during painful procedures.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Yakson touch — Yakson touch method will be started 5 minutes before the endotracheal aspiration procedure and continued until the completion of the procedure.The Yakson method continued for 15 minutes with steady touch (5 minutes), compassionate caressing (5 minutes), and repetition of steady touch (5 minutes).
  Arms: Yakson touch
Other: Gentle Human Touch — Gentle Human Touch (GHT) method will be started 5 minutes before the endotracheal aspiration procedure and continued until the completion of the procedure.The GHT method continued for 15 minutes.
  Arms: Gentle Human Touch
Other: Routine care — Infants in the Routine care will be applied swaddling. It will be started 5 minutes before the endotracheal aspiration procedure and continued until the completion of the procedure.
  Arms: Routine Care

SUMMARY:
The purpose of this study was to determine the effect of gentle human touch (GHT) and Yakson methods during endotracheal suctioning on pain, comfort and physiologic parameters response in preterm infants.

DETAILED DESCRIPTION:
Background: Preterm infants in the neonatal intensive care unit are exposed to various painful procedures, so different non-pharmacological pain control techniques are used to alleviate pain.

Aims: To determine the effect of gentle human touch (GHT) and Yakson methods during endotracheal suctioning on pain, comfort and physiologic parameters response in preterm infants.

Design: A randomized controlled crossover trial. Setting: This study was conducted in the neonatal intensive care unit between July 2022 and June 2023.

Methods: Thirty neonates were enrolled in this study based on inclusion criteria. The samples were randomly received a sequence of suctioning with Yakson and GHT and routine care. Neonatal Pain Agitation and Sedation Scale and COMFORT neo were used to collect the data.

ELIGIBILITY:
Inclusion Criteria:

* Infants in the 26-36/6 gestational week and at appropriate gestational age (AGA)
* Infants undergoing ventilator support with an endotracheal tube

Exclusion Criteria:

* Infants taking opiates and sedatives within four hours, having undergone a painful procedure at least one hour before
* Infants congenital anomalies, sepsis or haemorrhagic disease that might prevent Yakson and GHT
* Infants who underwent surgery and had a chest tube
* Infants with intracranial hemorrhage

Ages: 26 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Neonatal Pain Agitation and Sedation Scale (N-PASS) | Pain was assessed 1 minute before endotracheal aspiration, during endotracheal aspiration and 5 minutes after the endotracheal aspiration procedure.
  Pain will be evaluated using the Neonatal Pain Agitation and Sedation Scale (N-PASS).This scale was developed by Hummel Puchalski in 2000 for preterm and term babies. The Turkish validity and reliability study was conducted by Açıkgöz et al. in 2017. Crying, irritability, behavior-state, facial expression, extremity tone, and vital signs parameters are evaluated in the N-PASS scale. In this scale is evaluated with triple likert type and pain score can be between "0" and "10". Permission was obtained from the authors to use the scale.
Change in Oxygen saturation | Oxygen saturation was assessed 1 minute before endotracheal aspiration, during endotracheal aspiration and 5 minutes after the endotracheal aspiration procedure.
  Oxygen saturation of infants before, during, and after endotracheal aspiration were recorded to a computer using a Masimo Radical 7 Pulse Oximeter at 2-second intervals.
Change in Heart rate | Heart rate was assessed 1 minute before endotracheal aspiration, during endotracheal aspiration and 5 minutes after the endotracheal aspiration procedure.
  Heart rate of infants before, during, and after endotracheal aspiration were recorded to a computer using a Masimo Radical 7 Pulse Oximeter at 2-second intervals.

SECONDARY OUTCOMES:
COMFORTneo Scale | Comfort was assessed 1 minute before endotracheal aspiration, during endotracheal aspiration and 5 minutes after the endotracheal aspiration procedure.
  This scale was developed by Van Dijk et al. in 2009 for preterm babies. The Turkish validity and reliability study was conducted by Kahraman et al. in 2014. It is a 5-point Likert type scale consisting of six parameters: alertness, calmness/agitation, respiratory response, crying, body movements, facial tension, and muscle tone. The lowest score that can be obtained from the scale is 6 and the highest score is 30. It is emphasized that if the total score of the scale is between 9-13, the baby is comfortable, if it is between 14-30, the baby is in pain or distress, the baby is uncomfortable and needs interventions to provide comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye Dur, PhD, Principal Investigator — Izmir Democracy University; Seda Caglar, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Izmir Democracy University, Karabağlar, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No